CLINICAL TRIAL: NCT07313579
Title: Observational Prospective Cohort Study on Hyperthermic Intraperitoneal Chemoperfusion (HIPEC) in Gastric Cancer
Brief Title: Hyperthermic Intraperitoneal Chemoperfusion (HIPEC) in Gastric Cancer
Acronym: G-PEC
Status: Recruiting | Type: Observational
Sponsor: Ukrainian Society of Clinical Oncology (Other)
Responsible Party: Principal Investigator, Oleksii Dobrzhanskiy, Physician, Ukrainian Society of Clinical Oncology
Other Study IDs: 24999/2025
Record Dates: First submitted 2025-12-08; First posted 2026-01-02 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Gastric Cancer (GC); HIPEC; Peritoneal Metastases From Gastric Cancer; Hyperthermic Intraperitoneal Chemoperfusion
Keywords: Gastric cancer; HIPEC; Hyperthermic Intraperitoneal Chemoperfusion; FLOT; Lymphadenectomy; Gastrointestinal Neoplasms; Digestive System Neoplasms; Gastrointestinal Diseases; Stomach Diseases; Stomach Neoplasms; Chemotherapy, Adjuvant; Combined Modality Therapy; Drug Therapy; Surgical Procedures
MeSH Terms: conditions — Stomach Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Gastrointestinal Diseases; Stomach Diseases | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prophylactic cohort (T4a/T4b/cyt+): The cohort consists of individuals undergoing gastrectomy along with HIPEC.
  Interventions: Procedure: curative-intent surgery + HIPEC
- Low PCI cohort (PCI<7): Patients with low PCI undergo curative surgery with cytoreduction of visually detected peritoneal nodules followed by HIPEC
  Interventions: Procedure: curative-intent surgery + HIPEC

INTERVENTIONS:
Procedure: curative-intent surgery + HIPEC — Participants enrolled in this study will undergo curative-intent gastrectomy for gastric cancer, immediately followed by Hyperthermic Intraperitoneal Chemotherapy (HIPEC) performed during the same operative session. Dosage of drugs: mitomycin C 15 mg/m2, cisplatin 75mg/m2. The procedure is conducted according to a standardized protocol in National Cancer Institute

SUMMARY:
The study investigates the outcomes of hyperthermic intraperitoneal chemoperfusion (HIPEC) in combination with curative-intent gastrectomy in resectable locally-advanced and limited-metastatic (low peritoneal cancer index) gastric cancer.

DETAILED DESCRIPTION:
Several recent studies showed that near-perfect curative-intent R0 surgical technique combined with systemic chemotherapy or even immunotherapy may not always be enough to eliminate microscopic deposits or eliminate peritoneal dissemination in locally advanced gastric cancer or low peritoneal cancer-index (PCI) tumors. The risk of peritoneal dissemination is especially high for T4 tumors, for those with cytologically positive peritoneal washings. Moreover, the risk of peritoneal relapse in low PCI tumors is remarkably high. Combination of surgery and intraperitoneal chemotherapy aims to minimise the risks of the aforementioned peritoneal progression. In the study investigators perform curative surgery followed by single dose of hyperthermic intraperitoneal chemotherapy (HIPEC).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80
2. Hystologicaly proven gastric adenocarcinoma
3. ECOG status 0-1
4. Written consent to participate in the study
5. Medically and technically operable gastric tumor
6. Only T4a or T4b tumours with any peritoneal cytology status
7. Cytologically positive peritoneal washings (cyt+) with any T and N criteria
8. Adequate haemopoetic, renal and hepatic function (Hb > 120, PLT > 150*10^9/l, ALT < 60, AST <40, total bilirubin < 21 µmol/l, Creatinine clearance (male - 90-140, female - 80-130 ml/min)

Exclusion Criteria:

1. Pregnancy/breastfeeding
2. ECOG status 2-4
3. Concomitant malignancy
4. Mitomycin and/or Cisplatin hypersensitivity
5. Uncontrollable chronic diseases
6. Patients with coexisting malignancy other than basal cell carcinoma of the skin within the last five years.
7. Presence of metastases other than regional or peritoneal (such as liver, lungs, bone, brain, distant lymph nodes)
8. History of allergic reactions associated with cisplatin and Mitomycin C
9. Patients with psychiatric illness/social situations with impaired compliance
10. •Refusal to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients receiving care at oncological centers in Ukraine who meet all predefined eligibility criteria for this study. Investigators include individuals with for which Gastrectomy+HIPEC is considered an accepted or potentially beneficial treatment option according to national and international clinical guidelines. Participants will be recruited from tertiary surgical oncology hospitals and specialized cancer institutes across Ukraine.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2035-12-01 (Estimated)

PRIMARY OUTCOMES:
Peritoneal recurrence rate | From enrolment up to 5 years of follow-up
  Number of patients developed peritoneal recurence

SECONDARY OUTCOMES:
Distant recurrence rate | Time from diagnosis up to 5 years of follow-up
  Time from diagnosis to distant reccurence
Intraperitoneal chemotherapy complications rate | 30 days after chemotherapy
  Complications rate assessed by Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0 (Grade from 1 to 5)
Postoperative complications rate | 30 days after surgery
  Complications rate assessed by Clavien-Dindo scale (Grade from 1 to 5)
5-years overall survival | From the time of diagnosis up to 5 years of follow-up
  5-years overall survival
5-years relapse-free survival rate | Time from diagnosis up to 5 years of follow-up
  5-years relapse-free survival rate
Treatment-related quality of life assessed by Quality Of Life Questionnaire C30 version 3.0 | 6 months after treatment completion
  Treatment-related quality of life assessed by Quality Of Life Questionnaire C30 version 3.0 (lower score means better outcomes, higher score means worse outcomes)
Treatment-related quality of life assessed by Quality of Life Questionnaire-Stomach | 6 months after treatment completion
  Treatment-related quality of life assessed by Quality of Life Questionnaire-Stomach (lower score means better outcomes, higher score means worse outcomes)

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Kyiv, Ukraine